CLINICAL TRIAL: NCT04262934
Title: Multicenter Randomized Study : Does Correction of 25 OH-VITAmin D With Cholecalciferol Supplementation Increase Muscle Strength in hemoDIALysis Patients?
Brief Title: Does Correction of 25 OH-VITAmin D With Cholecalciferol Supplementation Increase Muscle Strength in hemoDIALysis Patients?
Acronym: VITADIAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Phoceen de Nephrologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITADIAL
Record Dates: First submitted 2020-01-27; First posted 2020-02-10 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-03

CONDITIONS: hemoDIALysis Patients
Keywords: 25 OH-VITAmin D supplementation; muscle strength
MeSH Terms: interventions — Cholecalciferol; Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholecalciferol treatment (Experimental): Arm A : Cholecalciferol 100.000 UI - oral - every month
  Interventions: Drug: Cholecalciferol 100.000 UI administration
- No treatment (Active Comparator): Arm B : No vitamin D administration
  Interventions: Other: No vitamin D administration

INTERVENTIONS:
Drug: Cholecalciferol 100.000 UI administration — One oral Administration - Every month
  Arms: Cholecalciferol treatment
Other: No vitamin D administration — No vitamin D administration
  Arms: No treatment

SUMMARY:
Muscle strength decreases as renal failure progresses. Low muscle strength affects more than 50% of hemodialysis patients and leads to daily life activities impairment. In the general population, numerous studies have linked low 25OH-vitamin D (25OHD) concentrations to the loss of the muscle strength and low physical performances. Data on native vitamin D and muscle function are scarce in the chronic renal failure (CKD) population, but low 25OHD levels have been associated with poor muscle strength. In this protocol of an ongoing study named VITADIAL testing if cholecalciferol supplementation in hemodialysis patients with low 25OHD improve their muscle strength.

DETAILED DESCRIPTION:
Prospective open randomized French multicenter study. All patients will have 25OHD levels ≤50nmol/L at randomization. One group will receive 100 000 UI cholecalciferol once a month during 6 months, the other group will receive no treatment during 6 months.

In order to randomize patients with 25OHD ≤50nmol/L, supplemented patients will undergo a 3 months wash-out period renewable 3 times (maximum of 12 months wash-out) until 25OHD reaches a level≤50nmol/L.

The main objective of this study is to analyze if a 6 months period of oral cholecalciferol (i.e. native vitamin D) supplementation improves muscle strength of hemodialysis patients with low 25OHD vitamin D levels. Muscle strength will be assessed at 0, 3 and 6 months, by handgrip strength measured with a quantitative dynamometer.

Secondary objectives are 1) to analyze 25OHD plasma levels after vitamin D wash-out and/or supplementation, as well as factors associated with 25OHD lowering speed during wash-out and 2) to analyze if this supplementation improves patient's autonomy, reduces frailty risk and improves quality of life.

ELIGIBILITY:
* Inclusion Criteria:

  * under hemodialysis for more than 3 months
  * aged over 18 years-old
  * gave their consent
* Non-inclusion criteria :

  * non fluent French speaker
  * incapacity to provide consent or to answer questionnaires
  * pregnancy or breast feeding
  * cognitive impairment
  * bedridden or life expectancy <1 year
  * active cancer
  * uncontrolled hyperparathyroidism as defined by the K-DIGO (iPTH>9x normal laboratory maximal value), cinacalcet treatment or hypocalcemia <2.0 mmol/L or hypercalcemia >2.7mmol/L
  * past osteoporosis fracture
  * treatment with active vitamin D
  * unable to perform handgrip measurement
  * 25OHD>50nmol/L without vitamin D treatment
  * cholecalciferol intolerance or allergy
* Exclusion Criteria:

  * 25OHD>50nmol/L after 12 months wash-out
  * hypercalcemia >2.7mmol/L
  * hyperparathyroidism (iPTH>9x normal laboratory maximal value) during wash-out or after randomization if patient is in the no treatment group
  * hypoparathyroidism (iPTH<3x normal laboratory lower value) in a patient receiving cholecalciferol
  * cholecalciferol intolerance or allergy
  * death, renal transplantation
  * pregnancy
  * consent withdrawal
  * renal recuperation allowing hemodialysis to stop
  * unability to perform handgrip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2024-06-08 (Estimated); Study Completion 2024-06-08 (Estimated)

PRIMARY OUTCOMES:
Muscle strength evaluation after 6 months period after cholecalciferol or no vitamin D treatment | At 6 months after randomization
  Muscle strength will be assessed by handgrip strength measured with a quantitative dynamometer

SECONDARY OUTCOMES:
Patient's autonomy after 6 months period of oral cholecalciferol | At 6 months post randomization (for patients treated)
  Katz Index of Independence in Activities of Daily Living (ADL)
Patient's frailty risk after 6 months period of oral cholecalciferol | At 6 months post randomization (for patients treated)
  The Frail Non-Disabled (FiND) Questionnaire
Patient's quality of life after 6 months period of oral cholecalciferol | At 6 months post randomization (for patients treated)
  Kidney Disease Quality of Life (KDQOL-SFtm) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas BATAILLE, MD, Principal Investigator — Institut Phoceen de Nephrologie
Locations (1):
- Pedinielli, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bataille S, Pedinielli N, Carreno E, Prezelin-Reydit M, Chauveau P, Jean G, Robert T, Bobot M, Seret G, Jouve E, Lavainne F, Serveaux M, Vrigneaud L, Gentile S. VITADIAL "Does correction of 25 OH-VITAmin D with cholecalciferol supplementation increase muscle strength in hemoDIALysis patients?": study protocol for a randomized controlled trial. Trials. 2021 May 25;22(1):364. doi: 10.1186/s13063-021-05302-9. PMID 34034786
- See also: Institut Phocéen de Néphrologie — https://www.nephrologuemarseille.fr